CLINICAL TRIAL: NCT03480074
Title: Endoscopic Stapling Versus Suture Ligation of Dorsal Venous Complex During Robot-Assisted Laparoscopic Prostatectomy: A Randomized Prospective Study
Brief Title: Staple vs. Suture in Robotic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PID 211077
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Staple Ligation (Active Comparator): Arm 1: Staple Ligation
  Interventions: Procedure: Staple Ligation
- Selective Suture Ligation (Active Comparator): Arm 2: Selective Suture Ligation
  Interventions: Procedure: Selective Suture Ligation
- Single Suture Ligation (Active Comparator): Arm 3: Single Suture Ligation
  Interventions: Procedure: Single Suture Ligation

INTERVENTIONS:
Procedure: Staple Ligation — Using a stapler that staples the DVC and then cuts it.
  Arms: Staple Ligation
Procedure: Selective Suture Ligation — Suture the DVC, suspend it to the pubic bone, and then cut.
  Arms: Selective Suture Ligation
Procedure: Single Suture Ligation — Cut the DVC, then pinpoint a specific blood vessel needed to sew/suture.
  Arms: Single Suture Ligation

SUMMARY:
The purpose of the study is to compare the results of three standard of care surgical methods [stapling versus selective suture ligation (cut, then sew) versus single suture ligation (sew, then cut) of the dorsal venous complex (DVC)] during robotic prostate surgery to see which is better for the patient's recovery.

DETAILED DESCRIPTION:
The dorsal venous complex (DVC) lies on top of the prostate gland, and carries blood away from the penis. It has to be tied off, or ligated, to remove the prostate gland. The DVC lies very close to nerves that help men get and maintain erections. In addition, the DVC is close to muscles that control passing urine. How the DVC is handled during prostate surgery may result in cancer being left behind to grow and spread in the body. The purpose of this study is to compare the results of stapling versus selective suture ligation (cut, then sew) versus single suture ligation (sew, then cut) of the DVC during robotic prostate surgery to see which is better for the patient's recovery.

This research is being done because doctors do not know which of these three commonly-used methods is better to reduce blood loss and reduce the chance of cancer left behind during surgery, and regain urine control and improve erectile function after surgery. Doctors also do not know if these methods affect the prostate-specific antigen (PSA) level in the blood after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Males over 18 years of age
* Must be scheduled to undergo standard of care robot-assisted laparoscopic prostatectomy (RALP)
* Must sign informed consent to be randomized between the three surgical arms

Exclusion Criteria:

* Patient is unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate study, only males eligible.
Enrollment: 300 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Post-operative Continence Rates | 2 years
  The amount of time after surgery for a patient to regain continence (is no longer using pads).

SECONDARY OUTCOMES:
Post-operative Erectile Function | 2 years
  The amount of time after surgery for a patient to regain erectile function.

CONTACTS AND LOCATIONS:
Overall Officials: James Porter, MD, Principal Investigator — Swedish Medical Center
Locations (1):
- Swedish Medical Center, Seattle, Washington, United States